CLINICAL TRIAL: NCT00062257
Title: A Phase II Study of Irofulven as First Line Therapy in Recurrent or Metastatic Gastric Cancer
Brief Title: Irofulven in Treating Patients With Recurrent or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Therapeutics Research Group (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CTRG-G15/02; CDR0000304669 (Registry Identifier: PDQ (Physician Data Query)); NCI-6041
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2005-03

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irofulven, use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well irofulven works in treating patients with recurrent or metastatic gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with recurrent or metastatic gastric cancer treated with irofulven.
* Determine the toxicity profile of this drug in these patients.
* Determine the overall survival of patients treated with this drug.

OUTLINE: This is a non-randomized, open-label, multicenter study.

Patients receive irofulven IV over 30 minutes on days 1 and 8. Courses repeat every 3 weeks in the absence of disease progression, unacceptable toxicity, or static disease after 4 courses in the absence of clinical benefit.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within 5-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed gastric adenocarcinoma

  * Recurrent or metastatic disease
  * Adenocarcinoma of the gastroesophageal junction eligible provided the majority of tumor bulk is below the junction
* Measurable disease

  * At least 1 lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active disseminated intravascular coagulation

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN for patients with liver metastases)
* Alkaline phosphatase no greater than 5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to irofulven
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Must have central or peripherally inserted central catheter

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa

Chemotherapy

* No prior chemotherapy for recurrent or metastatic disease
* Prior adjuvant or neoadjuvant chemotherapy allowed provided disease relapsed more than 6 months after therapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational or commercial agents or therapies for the malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, Study Chair — Prince of Wales Hospital
Locations (6):
- Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Singapore (3):
  - Cancer Institute at National University Hospital, Singapore
  - Johns Hopkins - Singapore, Singapore
  - National Cancer Centre - Singapore, Singapore
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea